CLINICAL TRIAL: NCT03505203
Title: Sleep-Safe: a Strong African American Families Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Georgia (Other)
Collaborators: Augusta University (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Justin Lavner, Associate Professor, University of Georgia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20180320; R01DK112874 (NIH)
Record Dates: First submitted 2018-04-03; First posted 2018-04-23 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2022-10

CONDITIONS: Weight Gain
Keywords: Responsive parenting; Mother-child relations; Infant feeding; Infant sleeping; Infant obesity
MeSH Terms: conditions — Weight Gain; Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one of two conditions: (1) Sleep Soothe (responsive parenting), where parents are given information on how to respond to their baby's cues related to sleeping and fussiness, and (2) Sleep Safe (safety control), where parents are given information on a safe sleep environment, as well as other strategies they can use to keep their baby safe.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sleep Soothe (Experimental): An intervention in which parents are given information on how to respond to their baby's cues related to sleeping and fussiness.
  Interventions: Behavioral: Sleep Soothe
- Sleep Safe (Active Comparator): An intervention in which parents are given information on a safe sleep environment, as well as other strategies to keep baby safe
  Interventions: Behavioral: Sleep Safe

INTERVENTIONS:
Behavioral: Sleep Soothe — An intervention in which parents are given information on how to respond to their baby's cues related to sleeping and fussiness.
  Arms: Sleep Soothe
Behavioral: Sleep Safe — An intervention in which parents are given information on a safe sleep environment, as well as other strategies to keep baby safe.
  Arms: Sleep Safe

SUMMARY:
Rapid weight gain during infancy is a powerful, and potentially malleable, risk factor for later overweight and obesity, but limited research has examined the impact of promising interventions when applied to the groups most at risk for rapid weight gain in infancy. The present study examines whether providing mothers of newborns with responsive parenting guidance during the first weeks of life to promote infant sleep and soothing can reduce rapid weight gain for African American infants born in low SES contexts.

DETAILED DESCRIPTION:
The study design is a randomized controlled trial. This trial will deliver a responsive parenting intervention (Sleep Soothe) to provide information on how to soothe, how to distinguish hunger from other distress, how to promote self-soothing, and bedtime routines. The responsive parenting intervention will be compared to a safety control group (Sleep Safe). The programs will be delivered across 2 sessions at 3-weeks and 8-weeks postpartum. Both interventions and all data collection will be delivered in participants' homes. Assessments will be conducted in participants' homes at 1-week postpartum, 3 weeks postpartum, 8 weeks postpartum, and 16-weeks postpartum.

Three hundred African American infants and their mothers will be recruited from the mother/baby nursery at Augusta University Medical Center. A dedicated recruitment coordinator will have access to electronic medical records systems in order to pre-screen mothers and infants. The recruitment coordinator will approach those who match basic inclusion criteria and will deliver an approved verbal script to pre-screened mothers to determine interest in participation. Interested mothers will respond to remaining screening questions in order to confirm eligibility. Once enrollment criteria are satisfied, informed consent will be obtained from the infant's mother during her hospital stay. Mothers will also complete selected demographic information. Anthropometric measurements will be obtained on the infant, mother, and father (optional). After enrollment, families will be scheduled for a research visit at their home at 1 week postpartum.

At home visit 1 (7-10 days postpartum), mothers (and fathers, if interested) will complete questionnaire measures using Qualtrics. There will also be measurements of infant weight and length. Families will be randomized to condition following this visit.

At home visit 2 (3 weeks postpartum), families will receive either the responsive parenting intervention or the safety control intervention. They will complete brief questionnaires. Measures of infant, maternal, and paternal (optional) weight will be obtained.

At home visit 3 (8 weeks postpartum), families will receive either the second part of the responsive parenting intervention or the second part of the safety control intervention. They will complete brief questionnaires. Measures of infant, maternal, and (optional: paternal) weight will be obtained. Mothers will be provided with activity monitors for themselves and for their babies that will be picked up by study staff after 7 days' use.

At home visit 4 (16 weeks postpartum), mothers will complete questionnaire measures (fathers' participation is optional). Measures of maternal and paternal (optional) weight will be obtained, as will measures of infant weight, length, and head circumference.

We test the following specific aims:

Specific Aim 1: To assess the effects of responsive parenting, focused on infant sleep and soothing, on reducing rapid weight gain from 3 to 16 weeks among African American infants. We hypothesize that infants in the Sleep Soothe condition will gain weight more slowly compared to infants in the Sleep Safe condition and have lower weight outcomes (i.e., BMI z scores, weight-for-length z scores, weight-for-age z scores) at age 16 weeks.

Specific Aim 2: To assess effects of responsive parenting on parental and infant behaviors. We hypothesize that compared with parents in the Sleep Safe condition, parents in the Sleep Soothe condition will show increases in responsive parenting, parenting self-efficacy, and the use of alternatives to feeding to soothe (white noise, pacifier, etc.), and decreases in feeding to soothe. Over time, infants in this condition will have longer sleep bouts and fewer feedings.

Specific Aim 3: To examine moderation of intervention effects by individual and contextual factors.

ELIGIBILITY:
Inclusion Criteria:

1. Infant > 37 0/7 weeks gestational age, apparently healthy and without significant morbidity
2. Singleton infant
3. Nursery/NICU/maternity stay of 7 days or less
4. Mother at least 17 years of age
5. Mother self-identifies as African American
6. Mother is primiparous

Exclusion Criteria:

1. Non-English speaking
2. Infant birth weight <2500 grams
3. Presence of a congenital anomaly or neonatal physical or metabolic condition that significantly affects a newborn's feeding (e.g. cleft lip, cleft palate, metabolic disease)
4. Any major maternal morbidities, pre-existing condition that would affect postpartum care or her ability to care for her newborn (e.g., narcotic drug use: heroin, cocaine, meth, pain pills, etc; on chemotherapy; uncontrolled MS; uncontrolled depression causing social service contact).
5. Plan for newborn to be adopted
6. Plan to move from area within four months of delivery
7. Residence further than 75 miles from Augusta, GA

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2018-03-04 (Actual); Primary Completion 2021-07-05 (Actual); Study Completion 2021-07-05 (Actual)

PRIMARY OUTCOMES:
Change in infants' weight for age from 3 weeks to 16 weeks (conditional weight gain) | 3 weeks to 16 weeks
  Standardized residuals from the linear regression of weight for age at 16 weeks on weight for age at 3 weeks, with length for age at birth and 16 weeks and infant age at the 16-week assessment entered as covariates

SECONDARY OUTCOMES:
Change in infants' weight for age | 3 weeks to 16 weeks
  Growth curve models of change in infants' weight for age
Weight-for-age z scores | 16 weeks
  Weight-for-age z scores at 16 weeks
Weight-for-length z scores | 16 weeks
  Weight-for-length z scores at 16 weeks
Infant BMI z scores | 16 weeks
  BMI z scores at 16 weeks

OTHER OUTCOMES:
Maternal report of infant sleep at 8 weeks | 8 weeks
  Sleep duration and number of night awakenings using the Brief Infant Sleep Questionnaire (Sadeh, 2004)
Maternal report of infant sleep at 16 weeks | 16 weeks
  Sleep duration and number of night awakenings using the Brief Infant Sleep Questionnaire (Sadeh, 2004)
Maternal sleep actigraphy | 8 weeks postpartum
  7-day actigraphy data to assess mothers' sleep duration
Infant soothing at 8 weeks | 8 weeks
  Parents use feeding for reasons other than in response to hunger
Infant soothing at 16 weeks | 16 weeks
  Parents use feeding for reasons other than in response to hunger
Infant feeding frequency at 16 weeks | 16 weeks
  Feeding frequency, use of bottle feeding, and introduction of solids using Babies Need Feeding (Stifter et al., 2011)
Safe sleep practices | 16 weeks
  Frequency of sleep safety practices (Fowler et al., 2013)
Child safety practices | 16 weeks
  Child safety practices assessed using the Framingham Safety Survey (Hansen et al., 1996)
Infant eating behavior | 16 weeks
  Infant eating behavior using the Baby Eating Behavior Questionnaire (Llewellyn et al., 2011)
Parental self-efficacy at 8 weeks | 8 weeks
  Perceived parental self-efficacy at 8 weeks using total score from the Karitane Parenting Confidence Scale (Crncec, Barnett, & Matthey, 2008)
Parental self-efficacy at 16 weeks | 16 weeks
  Perceived parental self-efficacy at 16 weeks using total score from the Karitane Parenting Confidence Scale (Crncec, Barnett, & Matthey, 2008)
Maternal feeding practices and beliefs at 8 weeks | 8 weeks
  Maternal feeding beliefs and behaviors using the Infant Feeding Styles Questionnaire (Thompson et al., 2009)
Maternal feeding practices and beliefs at 16 weeks | 16 weeks
  Maternal feeding beliefs and behaviors using the Infant Feeding Styles Questionnaire (Thompson et al., 2009)
Maternal depressive symptoms at 8 weeks | 8 weeks
  Maternal depressive symptoms at 8 weeks using the CES-D (Radloff, 1977)
Maternal depressive symptoms at 16 weeks | 16 weeks
  Maternal depressive symptoms at 16 weeks using the CES-D (Radloff, 1977)
Family routines | 8 weeks
  Extent to which there is order and routine versus chaos and confusion in their home. Uses total score from the Confusion, Hubbub, and Order Scale (Matheny et al., 1995)

CONTACTS AND LOCATIONS:
Overall Officials: Justin A Lavner, Ph.D., Principal Investigator — University of Georgia
Locations (1):
- University of Georgia, Athens, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lavner JA, Hohman EE, Beach SRH, Stansfield BK, Savage JS. Effects of a Responsive Parenting Intervention Among Black Families on Infant Sleep: A Secondary Analysis of the Sleep SAAF Randomized Clinical Trial. JAMA Netw Open. 2023 Mar 1;6(3):e236276. doi: 10.1001/jamanetworkopen.2023.6276. PMID 37000448
- [Background] Hohman EE, Savage JS, Stansfield BK, Lavner JA. Sleep SAAF Responsive Parenting Intervention for Black Mothers Impacts Response to Infant Crying: A Randomized Clinical Trial. Acad Pediatr. 2024 Jan-Feb;24(1):97-104. doi: 10.1016/j.acap.2023.04.012. Epub 2023 May 5. PMID 37148966
- [Background] Hart AR, Beach SRH, Hart CN, Smith JJ, Stansfield BK, Lavner JA. Responsive parenting and Black mothers' postpartum sleep: Secondary analysis of a randomized controlled trial. Health Psychol. 2024 Jun;43(6):438-447. doi: 10.1037/hea0001363. Epub 2024 Feb 8. PMID 38330306
- [Background] Weber DM, Bryant CM, Williamson HC, Mussa K, Lavner JA. Predictors of change in relationship satisfaction among Black postpartum mothers. Fam Process. 2024 Jun;63(2):768-787. doi: 10.1111/famp.12990. Epub 2024 Mar 28. PMID 38548477
- [Background] Weber DM, Williamson HC, Bryant CM, Mussa KS, Lavner JA. Patterns and predictors of change in relationship status among Black mothers over 16 weeks postpartum. J Fam Psychol. 2024 Aug;38(5):751-762. doi: 10.1037/fam0001238. Epub 2024 Jun 17. PMID 38884990
- [Background] Adesogan O, Beach SRH, Carter SE, Metzger IW, Lavner JA. Effects of a responsive parenting intervention on Black mothers' depressive symptoms postpartum: Secondary analysis of a randomized clinical trial. J Consult Clin Psychol. 2024 Dec;92(12):828-835. doi: 10.1037/ccp0000926. PMID 39715425
- [Background] Moore AM, Smith JJ, Stansfield BK, Savage JS, Lavner JA. Patterns and Predictors of Breast Milk Feeding from Birth to Age 4 Months among Primiparous African American Mother-Infant Dyads. Nutrients. 2022 Jun 4;14(11):2350. doi: 10.3390/nu14112350. PMID 35684150
- [Background] Lavner JA, Savage JS, Stansfield BK, Beach SRH, Marini ME, Smith JJ, Sperr MC, Anderson TN, Hernandez E, Moore AM, Caldwell AL, Birch LL. Effects of the Sleep SAAF responsive parenting intervention on rapid infant weight gain: A randomized clinical trial of African American families. Appetite. 2022 Aug 1;175:106080. doi: 10.1016/j.appet.2022.106080. Epub 2022 May 13. PMID 35577176
- [Background] Hernandez E, Lavner JA, Moore AM, Stansfield BK, Beach SRH, Smith JJ, Savage JS. Sleep SAAF responsive parenting intervention improves mothers' feeding practices: a randomized controlled trial among African American mother-infant dyads. Int J Behav Nutr Phys Act. 2022 Oct 1;19(1):129. doi: 10.1186/s12966-022-01366-1. PMID 36183135
- [Background] Lavner JA, Stansfield BK, Beach SRH, Brody GH, Birch LL. Sleep SAAF: a responsive parenting intervention to prevent excessive weight gain and obesity among African American infants. BMC Pediatr. 2019 Jul 5;19(1):224. doi: 10.1186/s12887-019-1583-7. PMID 31277694
- [Derived] Hart AR, Beach SRH, Hart CN, Metzger IW, Lavner JA. Effects of contextual stress on Black mothers' self-reported and actigraph-estimated postpartum sleep. Sleep. 2025 Jul 11;48(7):zsaf023. doi: 10.1093/sleep/zsaf023. PMID 40036969